CLINICAL TRIAL: NCT01684475
Title: A STUDY TO EVALUATE THE EFFICACY OF CJH1 [CLR4001] IN THE TREATMENT OF PARKINSON'S DISEASE
Brief Title: A STUDY TO EVALUATE THE EFFICACY OF CJH1 (CLR4001) IN PARKINSON'S DISEASE
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandra Marine and General Hospital (Other)
Responsible Party: Principal Investigator, Craig Hudson MD, Psychiatrist, Alexandra Marine and General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: CJH1 Trial
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Parkinson's Disease
Keywords: Novel Treatment Parkinson's disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with CJH1 (Experimental)
  Interventions: Drug: CJH1 (CLR4001)

INTERVENTIONS:
Drug: CJH1 (CLR4001)

SUMMARY:
The purpose of this study is to assess the ability of CJH1 to increase the sensitivity of dopamine receptors and thereby reduce symptoms of Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Patient's with Parkinson's disease

Exclusion Criteria:

* Contraindications to study medication

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-09; Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Reduced signs and symptoms of Parkinson's disease | 8 weeks
  Reduced signs and symptoms of Parkinson's disease

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Rural Health Research, Goderich, Ontario, Canada